CLINICAL TRIAL: NCT03059719
Title: A Randomized, Open, Comparative to the Positive-Controlled, Parallel Group, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PB-119 to Subjects Newly Diagnosed as Type 2 Diabetes Mellitus
Brief Title: Clinical Trial for PB-119 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICP-I-2015-01
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Type II Diabetes Mellitus
Keywords: safety; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PB-119 injection (Experimental): PB119 injection 25ug or 50ug once each week, for three months
  Interventions: Biological: PB-119 injection
- Exenatide Injection (Byetta) (Active Comparator): Byetta 5ug or 10ug twice each day, for three months
  Interventions: Biological: Exenatide injection(Byetta)

INTERVENTIONS:
Biological: Exenatide injection(Byetta)
  Arms: Exenatide Injection (Byetta)
Biological: PB-119 injection
  Arms: PB-119 injection

SUMMARY:
This is a randomized, opened, positive drug-controlled (Exenatide, Byetta), sequential parallel group, multiple dose study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of twelve once-weekly subcutaneous doses of PB-119 to subjects with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
There are two study phases according to different doses of investigational drug Phase 1：1 investigational group and 1 control group, i.e.; investigational drug PB-119 injection 25µg group and control drug exenatide group.

Phase 1： Plan to have 1 or 2 investigational group according to the study result from phase 1, i.e., investigational drug PB-119 injection 50 µg group and control drug exenatide group.

Subject Number：18 subjects will be randomized to each group, with equal number of females and males. 12 subjects will be in PB-119 group, 6 subjects will be in exenatide group.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects between the ages of 18~45 (inclusive) years, the ratio of females to males is approximately 1:1;
2. Subject has been disguised as type 2 diabetes within 5 years of screening, and met the diagnosis criteria of type 2 diabetes in guidance from WHO and Chinese Diabetes Society (CDS);
3. Subject didn't received any treatment for diabetes before screening, subject has been on diet control for more than 3 months, Fasting Plasma Glucose (FPG) was 7.0 ~ 13.0 mmol / L (including boundary value), and the glycosylated hemoglobin (HbA1c) was 7.0% ~ 10% (Including boundary values);
4. Female weight of ≥45 kg, male weight of ≥50 kg, subject body mass index (BMI) between 19~30 kg/m2 (inclusive);
5. Subject can understand the procedures and methods of this clinical trial, is willing to participate and sign the written informed consent;

Exclusion Criteria:

1. Subject was diagnosed as type 1 diabetes
2. Subject has acute complications of diabetes, such as ketoacidosis or hyperosmolar coma within 6 months before screening;
3. Subject who is allergic to exenatide, investigational drug or any ingredients (citric acid, mannitol, m-cresol); or have specific severe drug allergy history
4. Patient has specific cardiovascular disease, such as unstable angina pectoris, myocardial infarction, hypertension with poor control using one antihypertensive drugs (mean sitting systolic blood pressure ≥ 160mmHg or diastolic blood pressure ≥ 95mmHg), severe arrhythmia, QTc Prolonged, cardiac dysfunction and so on;
5. Subject who has liver and kidney dysfunction (ALT or AST> 2 times of upper limit of normal reference range, or TBIL> 1.5 times of upper limit of normal reference range, or Cr> upper limit of normal reference range);
6. Subject who's triglyceride≥5mmol/L；
7. Subject who has acute or chronic hepatitis, or other liver disease
8. Known medical history of acute pancreatitis or chronic pancreatitis, or pancreatic amylase> upper limit of normal reference range, or serum lipase> upper limit of normal reference range;
9. Subject has disease which may impact gastric emptying, such as gastroparesis, gastric outlet obstruction, intestinal obstruction, or received gastric bypass surgery, or long-term use of drugs which may have direct impact on gastrointestinal peristalsis;
10. Subject has any clinical significant major disease history or medical history of respiratory system, digestive system, nervous system, hematology system, urology system, immunology, psychiatric system and metabolic disorders etc.
11. Subject has liver, kidney or gastrointestinal partial resection surgery
12. Subject has drug abuse or alcoholic
13. Subject who has received any Chinese and western medication treatment for diabetes;
14. Subject who has taken any prescription or over-the-counter medications (such as orlistat, sibutramine, rimonabant, phenylpropanol or chlorpheniramine) that promote weight loss within 3 months before study;
15. Take any medications that may affect test results, such as antibiotics, non-steroidal anti-inflammatory drugs, antacids containing aluminum or magnesium, diuretics, anticoagulants, central nervous system inhibitors, systemic corticosteroids, medications to slow down the gastrointestinal motility, and any drug that may possibly affect the absorption of the drug within 2 weeks before screening;
16. Participated any clinical trial within 3 months before trial;
17. Female who is pregnant or lactating;
18. Subject who is not able to use contraceptive methods that is medically recognized during study;
19. Subject who cannot complete study due to other reason or determined by investigators as inappropriate to participate this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-10-27 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AE (safety and tolerability) | the change form base line lab values at 3 months
  N of participants with abnormal lab values and AE relevant to the treatment

SECONDARY OUTCOMES:
PB-119 blood concentration | hour0, hour12, hour24, hour48, hour72, hour96, hour120, hour144, hour168, hour336, hour504, hour672, hour1344, hour1848, hour1872, hour1896, hour1920, hour2016, hour2112, hour2184 and hour2580
  N of PB-119 blood concentration

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Lv, Principal Investigator — No.1 Hospital of Peking University
Locations (1):
- No.1 Hospital of Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No